CLINICAL TRIAL: NCT01688076
Title: Treatment of Forehead/Glabellar Rhytide Complex With Botulinum Toxin A Injection: Impact of Muscle Contraction on Onset of Action, Efficacy, and Duration of Treatment
Brief Title: Treatment of Forehead/Glabellar Rhytide Complex With Botulinum Toxin A Injection
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology - Head and Neck Surgery, and Surgery-Organ Transplantation, Northwestern University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STU56722
Record Dates: First submitted 2012-04-04; First posted 2012-09-19 (Estimated); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Forehead Rhytid Complex; Glabellar Rhytid Complex
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Muscle contractions (Experimental): Under supervision by study personnel, subjects be asked to make active muscle contractions for one hour after Botox injections. Subjects will return for follow-up visits.
  Interventions: Procedure: Botulinum Toxin A
- No muscle contractions (Active Comparator): Patients will be asked to not perform muscle contractions following Botox injections.
  Interventions: Procedure: Botulinum Toxin A

INTERVENTIONS:
Procedure: Botulinum Toxin A — Forehead will be injected with Botox.

SUMMARY:
This cross-over design study will evaluate the onset of action, efficacy, and duration of botulinum toxin A treatment on forehead/glabellar rhytid complexes with and without subsequent muscle contraction.

DETAILED DESCRIPTION:
In this cross-over design study, the investigators will evaluate whether active muscle contraction following Botox® injection of the forehead/glabellar rhytid complex will impact the onset of action, efficacy, and duration of Botox® treatment.

ELIGIBILITY:
Inclusion Criteria:

* In good health
* Is 18-65 years of age
* Has static and dynamic forehead/glabellar wrinkles
* Has decided to receive Botox® treatment for their forehead/glabellar wrinkles
* Has the willingness and ability to understand and provide informed consent and communicate with the investigator
* Is willing to return for follow-up visits

Exclusion Criteria:

* Pregnant or lactating
* Has received the following treatments in the forehead or glabellar region:

  * botulinum toxin injections in the past 6 months
  * ablative laser procedure in the past 6 months
  * radiofrequency device treatment in the past 6 months
  * ultrasound device treatment in the past 6 months
  * medium to deep chemical peel in the past 6 months
  * temporary soft tissue augmentation material in the past year
  * semi-permanent soft tissue augmentation material in the past 2 years
  * permanent soft tissue augmentation material
* Is planning to receive within the next year, any cosmetic procedure (such as any chemical peels, botulinum toxin injections, ablative or non-ablative laser procedures, filler injections, radiofrequency procedures, dermabrasion, ultrasound and face lifting procedures) in the forehead or glabellar region.
* Is planning to use tretinoin or retinoic acid in the next year
* Has an active infection in the forehead or glabellar region (excluding mild acne)
* Is allergic to cow's-milk protein
* Is allergic to albumin
* Taking aminoglycoside
* Is currently using anticoagulation therapy
* Has a history of bleeding disorders
* Is unable to understand the protocol or to give informed consent
* Is unable to return for follow-up visits
* Has a mental illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-01; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of Forehead Wrinkles with Honeck Four Point Rating Scale | 13 months
  A single dermatologist will rate each photograph of the subject's forehead/glabellar rhytid complex at baseline, 1 day, 2 days, 3 days, 4 days, 7 days, 2 weeks, 7 months and 1 day, 7 months and 2 days, 7 months and 3 days, 7 months and 4 days, 7 months and 7 days, and 7 months and 2 weeks. A glabellar wrinkle score and a forehead wrinkle score will be assigned to each photograph. The dermatologist will not know at what point in time the photographs were taken.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | 13 months
  Side effects and adverse events will be assessed
Level of Satisfaction | 7 months
  Patients will be asked to rate their satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States